CLINICAL TRIAL: NCT04199819
Title: The Use of Novel Hepatitis B Virus (HBV) Biomarkers to Detect Occult HBV Infection in Liver Donors Positive for Antibody to Hepatitis B Core Antigen (Anti-HBc) in Liver Transplantation
Brief Title: Detecting Occult HBV Infection in Liver Donors Positive for Antibody to Hepatitis B Core Antigen (Anti-HBc)
Acronym: OBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Yan Yue Fung, Principal Investigator, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: occult HBV infection 01
Record Dates: First submitted 2019-12-03; First posted 2019-12-16 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Occult Hepatitis B; Liver Transplant; Complications
Keywords: occult hepatitis b; liver transplantation; novel biomarkers
MeSH Terms: interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HBsAg-negative recipients (Other): Recipients who are HBsAg-negative will undergo a panel of test to detect HBV viral markers. In addition, real-time PCR will be used to determine the presence of intrahepatic HBV DNA and cccDNA on the explant histology. Patients with evidence of OBI, as characterized by any one positive biomarker (serum HBV DNA, serum HBV RNA, serum HBcrAg, intrahepatic HBV DNA, intrahepatic cccDNA) in either the donor or recipient, will be commenced on life-long oral nucleos(t)ide analog therapy as part of their routine antiviral prophylaxis. For those without evidence of OBI, that is, negative for all biomarkers, no antiviral prophylaxis will be given.
  Interventions: Drug: entecavir

INTERVENTIONS:
Drug: entecavir — Patients with evidence of OBI, as characterized by any one positive biomarker (serum HBV DNA, serum HBV RNA, serum HBcrAg, intrahepatic HBV DNA, intrahepatic cccDNA) in either the donor or recipient, will be commenced on life-long oral nucleos(t)ide analog therapy as part of their routine antiviral prophylaxis.
  Other Names: antiviral therapy

SUMMARY:
After LT, long-term immunosuppressive therapy is required to prevent organ rejection. Therefore, for organs which may harbour OBI, there is a risk of reactivation which may result in liver graft failure. As a consequence, all patients who receive an anti-HBc positive graft will receive antiviral prophylaxis. Currently, all such patients will be commenced on life-long entecavir, which is highly effective in preventing reactivation.2 One major disadvantage of using such a blanket approach is that a significant proportion of anti-HBc donors may not actually have underlying occult HBV infection, and recipients of such grafts may not require lifelong antiviral therapy. Current markers such as HBsAg and HBV DNA are not sensitive enough to detect the presence of OBI.

This is the first trial proposed to look at the efficacy of these novel HBV biomarkers in identifying occult HBV infection when used in combination, and to identify patients who will not need long term antiviral prophylaxis.

DETAILED DESCRIPTION:
Liver transplantation (LT) is potential curative for those with liver failure or hepatocellular carcinoma. In Hong Kong, where HBV infection remains endemic, chronic HBV (CHB) infection remains the leading indication for LT. Due to the low rate of organ donation, hepatitis B surface antigen (HBsAg) negative donors who are anti-HBc positive are frequently used. There is potential for anti-HBc positive donors to harbor OBI, defined as the presence of liver and/or serum HBV DNA without serological evidence of chronic infection (HBsAg negative).1 Hence, there is a risk of transmitting HBV infection when these grafts are transplanted to HBsAg negative recipients (de novo HBV infection). Nonetheless, anti-HBc positive donors represent an important source of organs in HBV endemic area, including Hong Kong, with a high prevalence rate (37%) of HBsAg negative but anti-HBc positive population.

After LT, long-term immunosuppressive therapy is required to prevent organ rejection. Therefore, for organs which may harbour OBI, there is a risk of reactivation which may result in liver graft failure. As a consequence, all patients who receive an anti-HBc positive graft will receive antiviral prophylaxis. Currently, all such patients will be commenced on life-long entecavir, which is highly effective in preventing reactivation.2 One major disadvantage of using such a blanket approach is that a significant proportion of anti-HBc donors may not actually have underlying occult HBV infection, and recipients of such grafts may not require lifelong antiviral therapy. Current markers such as HBsAg and HBV DNA are not sensitive enough to detect the presence of OBI.

More recently a panel of novel HBV biomarkers have emerged.3,4 These include quantification of anti-HBc, HBV RNA, hepatitis B core-related antigen (HBcrAg), and intrahepatic covalently closed circular DNA (cccDNA) levels. Some of these markers have been associated with OBI, and may predict HBV reactivation for immunosuppressed patients.5,6

This is the first trial proposed to look at the efficacy of these novel HBV biomarkers in identifying occult HBV infection when used in combination, and to identify patients who will not need long term antiviral prophylaxis

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient age ≥18 years undergoing liver transplantation
* 2. Donor HBsAg- and anti-HBc+

Exclusion Criteria:

* 1. Recipient of multiple solid organ transplants
* 2. Patient undergoing re-transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of HBsAg-negative recipients of an anti-HBc+ graft needing antiviral therapy | 2 years
  Proportion of HBsAg-negative recipients of an anti-HBc+ graft needing antiviral therapy

SECONDARY OUTCOMES:
Prevalence of occult hepatitis B infection in HBsAg-/anti-HBc+ donors | 2 years
  Prevalence of occult hepatitis B infection in HBsAg-/anti-HBc+ donors

CONTACTS AND LOCATIONS:
Overall Officials: James Fung, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong